CLINICAL TRIAL: NCT05836740
Title: Efficacy and Safety of Minocycline in Patients With Moderate to Severe Acute Ischemic Stroke: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase III Trial
Brief Title: Efficacy and Safety of Minocycline in Patients With Moderate to Severe Acute Ischemic Stroke
Acronym: EMPHASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2023-007-01
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Minocycline
MeSH Terms: conditions — Ischemic Stroke; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: This trial was a prospective, randomized, multicenter, double-blind, placebo-controlled parallel trial. Participants were randomly assigned according to the ratio of the experimental group: control group =1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Minocycline drug used in the study is indistinguishable from the Minocycline placebo (the shape, color, and appearance are identical).
  In addition, to ensure the blind method, the drug packaging and batch numbers of the two groups are identical, and the packaging batch numbers are uniformly marked.
  During the implementation of the study, except for the authorized personnel of the company's supply chain, research management department, and subject security department, members of each research execution group, research center personnel, and CRO data processing personnel cannot view the randomization scheme. The blind method was also used to evaluate the outcome. The participants were randomly divided into groups and blinded to the members of the adjudication committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline treatment group (Active Comparator): Minocycline Hydrochloride Capsules (50 mg per capsule) The first dose should be given immediately after randomization (within 30 minutes); 200mg (4 capsules) for the first dose; Subsequently, 100mg (2 capsules) will be administered once every 12 hours, a total of 9 times (lasting 4.5 days; the subject with dysphagia will be administrated through a nasal feeding tube)
  Interventions: Drug: Minocycline hydrochloride capsule
- Minocycline placebo-control group (Placebo Comparator): Placebo of Minocycline Hydrochloride capsules (50mg per capsule, containing 0 mg of Minocycline) The method of administration was the same as that of treatment group.
  Interventions: Drug: Placebo capsules of Minocycline hydrochloride capsules

INTERVENTIONS:
Drug: Minocycline hydrochloride capsule — 50 mg per capsule, containing 50mg of Minocycline Hydrochloride.
  Arms: Minocycline treatment group
Drug: Placebo capsules of Minocycline hydrochloride capsules — 50 mg per capsule, containing 0mg of Minocycline Hydrochloride.
  Arms: Minocycline placebo-control group

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of Minocycline versus placebo in the treatment of patients with moderate to severe acute ischemic stroke.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of 4.5-days Minocycline versus placebo in patients with moderate to severe acute ischemic stroke within 72 hours of onset. In addition, we will explore the effect of Minocycline versus placebo on indicators of venous neuroinflammation and thrombo-inflammation at different time points in patients with moderate to severe acute ischemic stroke within 72 hours of onset.

The primary objective is to evaluate the effect of Minocycline in improving the level of mRS score to 0-1 in patients with moderate to severe acute ischemic stroke within 72 hours of onset.

The trial was divided into three phases: screening/baseline period, treatment period, and follow-up period. The visit schedule is as follows: Randomized participants were interviewed at screening/baseline period, 24±2 hours, 6±1 days, 90±7 days after randomization, and when events occurred.

ELIGIBILITY:
Inclusion criteria:

1. 18≤Age≤80 years old;
2. Patients with acute ischemic stroke confirmed by CT or MRI within 72 hours of onset;
3. 4≤NIHSS≤25, and Ia≤1;
4. First stroke or mRS 0-1 before the onset of current stroke;
5. Patients or his/her legal representatives are able to understand and sign the informed consent.

Exclusion criteria:

1. History of pseudomembranous colitis or antibiotic-related colitis.
2. Allergic to tetracycline antibiotics or any component of the investigational drug.
3. Known to be resistant to other tetracyclines.
4. Took tetracycline antibiotics within previous one week.
5. Known community-acquired bacterial infection, such as pneumonia or urinary tract infection.
6. History of intracranial hemorrhagic diseases within previous 3 months, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/external hematoma, etc.
7. Intracranial tumors, vascular malformations and other intracranial space-occupying lesions.
8. Rare or unknown etiology of LVO, such as dissection and vasculitis.
9. Severe hepatic insufficiency, renal insufficiency or receiving dialysis before randomization for various reasons (Severe hepatic insufficiency was defined as ALT >3 times the upper limit of normal value or AST >3 times the upper limit of normal value; Severe renal insufficiency was defined as creatinine > 3.0 mg/dl [265.2 μmol/L] or glomerular filtration rate<30 ml/min/1.73m2).
10. Bleeding tendency (including but not limited to): platelet count <100×109/L; Administration of oral warfarin and INR>2; Administration of heparin within previous 48 hours and APTT≥35s; Hereditary bleeding disorders, such as hemophilia.
11. Received any of the following treatments within previous 3 months: systemic retinoic acid, androgen/antiandrogen therapy (e.g., anabolic steroids, andiolactone).
12. History of intracranial or spinal surgery within previous 3 months; History of therapeutical surgery or major physical trauma within previous 1 month.
13. Women of childbearing age who do not use effective contraception and have no negative pregnancy test records; Women during lactation and pregnancy.
14. Life expectancy of less than 6 months due to advanced stage of comorbidity.
15. Participated in other interventional clinical trials within previous 3 months.
16. Other conditions that are not suitable for participating in this clinical trial, such as inability to understand and/or follow the research procedures due to mental, cognitive, emotional, or physical disorders, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1724 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
mRS score 0-1 | At 90±7 days after randomization.
  Modified Rankin Scale score.

SECONDARY OUTCOMES:
mRS score. | At 90±7 days after randomization.
  Modified Rankin Scale score.
Changes in NIHSS score compared with baseline score. | At 24±1 hours and 6±1 days after randomization.
  NIHSS score
Changes in hs-CRP level compared with baseline level. | At 6±1 days after randomization.
  hs-CRP was examined to evaluate the level of systematic inflammation
Early neurological deterioration. | At 24±2 hours and 6±1 days after randomization.
  Early neurological deterioration was defined as any new neurological symptoms or signs that occur within several hours or days of onset, as well as the progression of existing neurological deficit symptoms or signs.
Recurrent stroke. | At 90±7 days after randomization.
  Recurrent stroke includes recurrent ischemic stroke and recurrent hemorrhagic stroke.
Recurrent ischemic stroke. | At 90±7 days after randomization.
  The condition of recurrent ischemic stroke.
Combined vascular events. | At 90±7 days after randomization.
  Combined vascular events referred to stroke, myocardial infarction, and vascular death.
Quality of life (EQ-5D) score. | At 90±7 days after randomization.
  Scores of EuroQol (Quality of life) -5 Dimensions.

OTHER OUTCOMES:
Changes in the levels of venous neuroinflammation indicators and thrombotic inflammation indicators compared with baseline levels. | At 24±2 hours and 6±1 days after randomization.
  Venous neuroinflammation indicators (NF-L, S100B, copeptin, etc.) and thrombotic inflammation indicators (plasma sGPVI, sADAMTS 13, sCD40L, sP-selectin, etc.)
Cerebral hemodynamic function. | At 6±1 days and 90±7 days after randomization.
  Cerebral hemodynamics was reflected by cerebral autoregulation function, and autonomic nervous function was evaluated by heart rate variability.
Changes in the levels of venous intestinal flora metabolites compared with baseline levels | At 6±1 days after randomization.
  plasma TMAO and its precursors, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD+MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (58):
- China (58):
  - The Eighth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Chongqing Donghua Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Shenzhen Hospital, Southern Medical University, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - The Sixth People's Hospital of Hengshui, Hengshui, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Dengzhou People's Hospital, Dengzhou, Henan
  - Xiuwu People's Hospital, Jiaozuo, Henan
  - Jiyuan Chinese Medical Hospital, Jiyuan, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Mengjin People's Hospital, Luoyang, Henan
  - Luoning People's Hospital, Luoyang, Henan
  - Mengzhou People's Hospital, Mengzhou, Henan
  - Nanle Zhongxing Hospital, Puyang, Henan
  - Sui Chinese Medical Hospital, Shangqiu, Henan
  - Xingyang People's Hospital, Zhengzhou, Henan
  - Biyang People's Hospital, Zhumadian, Henan
  - Pingyu People's Hospital, Zhumadian, Henan
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Shimen People's Hospital, Changde, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First People's Hospital of Chenzhou/The First Affiliated Hospital of Xiangnan University, Chenzhou, Hunan
  - Hengyang Central Hospital, Hengyang, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Changzhou Wujin Traditional Chinese Medicine Hospital, Changzhou, Jiangsu
  - Rudong People's Hospital, Nantong, Jiangsu
  - The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Benxi Central Hospital, Benxi, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng Central Hospital, Liaocheng, Shandong
  - The Third People's Hospital of Liaocheng, Liaocheng, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanghai Pudong New Area Gongli Hospital, Shanghai, Shanghai Municipality
  - Xi'an International Medical Center Hospital, Xi'an, Shannxi
  - Yuci District People's Hospital, Jinzhong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Production and Construction Corps 13 Division Red Star Hospital, Hami, Xinjiang
  - Xinjiang Production&Construction Corps Hospital, Ürümqi, Xinjiang
  - Affiliated Hangzhou First People's Hospital, Westlake University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Tiantan Hospital, Beijing
  - Ningjin People's Hospital, Dezhou
  - Zouping City People's Hospital, Jining

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou M, Wang H, Zhu J, Chen W, Wang L, Liu S, Li Y, Wang L, Liu Y, Yin P, Liu J, Yu S, Tan F, Barber RM, Coates MM, Dicker D, Fraser M, Gonzalez-Medina D, Hamavid H, Hao Y, Hu G, Jiang G, Kan H, Lopez AD, Phillips MR, She J, Vos T, Wan X, Xu G, Yan LL, Yu C, Zhao Y, Zheng Y, Zou X, Naghavi M, Wang Y, Murray CJ, Yang G, Liang X. Cause-specific mortality for 240 causes in China during 1990-2013: a systematic subnational analysis for the Global Burden of Disease Study 2013. Lancet. 2016 Jan 16;387(10015):251-72. doi: 10.1016/S0140-6736(15)00551-6. Epub 2015 Oct 26. PMID 26510778
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Result] Wardlaw JM, Murray V, Berge E, del Zoppo G, Sandercock P, Lindley RL, Cohen G. Recombinant tissue plasminogen activator for acute ischaemic stroke: an updated systematic review and meta-analysis. Lancet. 2012 Jun 23;379(9834):2364-72. doi: 10.1016/S0140-6736(12)60738-7. Epub 2012 May 23. PMID 22632907
- [Result] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Result] Tao C, Nogueira RG, Zhu Y, Sun J, Han H, Yuan G, Wen C, Zhou P, Chen W, Zeng G, Li Y, Ma Z, Yu C, Su J, Zhou Z, Chen Z, Liao G, Sun Y, Ren Y, Zhang H, Chen J, Yue X, Xiao G, Wang L, Liu R, Liu W, Liu Y, Wang L, Zhang C, Liu T, Song J, Li R, Xu P, Yin Y, Wang G, Baxter B, Qureshi AI, Liu X, Hu W; ATTENTION Investigators. Trial of Endovascular Treatment of Acute Basilar-Artery Occlusion. N Engl J Med. 2022 Oct 13;387(15):1361-1372. doi: 10.1056/NEJMoa2206317. PMID 36239644
- [Result] Shi K, Tian DC, Li ZG, Ducruet AF, Lawton MT, Shi FD. Global brain inflammation in stroke. Lancet Neurol. 2019 Nov;18(11):1058-1066. doi: 10.1016/S1474-4422(19)30078-X. Epub 2019 Jul 8. PMID 31296369
- [Result] Yang JL, Yang YR, Chen SD. The potential of drug repurposing combined with reperfusion therapy in cerebral ischemic stroke: A supplementary strategy to endovascular thrombectomy. Life Sci. 2019 Nov 1;236:116889. doi: 10.1016/j.lfs.2019.116889. Epub 2019 Oct 11. PMID 31610199
- [Result] McGarry T, Biniecka M, Veale DJ, Fearon U. Hypoxia, oxidative stress and inflammation. Free Radic Biol Med. 2018 Sep;125:15-24. doi: 10.1016/j.freeradbiomed.2018.03.042. Epub 2018 Mar 27. PMID 29601945
- [Result] Stoll G, Nieswandt B. Thrombo-inflammation in acute ischaemic stroke - implications for treatment. Nat Rev Neurol. 2019 Aug;15(8):473-481. doi: 10.1038/s41582-019-0221-1. Epub 2019 Jul 1. PMID 31263257
- [Result] Kollikowski AM, Schuhmann MK, Nieswandt B, Mullges W, Stoll G, Pham M. Local Leukocyte Invasion during Hyperacute Human Ischemic Stroke. Ann Neurol. 2020 Mar;87(3):466-479. doi: 10.1002/ana.25665. Epub 2020 Jan 16. PMID 31899551
- [Result] El Amki M, Wegener S. Improving Cerebral Blood Flow after Arterial Recanalization: A Novel Therapeutic Strategy in Stroke. Int J Mol Sci. 2017 Dec 9;18(12):2669. doi: 10.3390/ijms18122669. PMID 29232823
- [Result] Bustamante A, Ning M, Garcia-Berrocoso T, Penalba A, Boada C, Simats A, Pagola J, Ribo M, Molina C, Lo E, Montaner J. Usefulness of ADAMTS13 to predict response to recanalization therapies in acute ischemic stroke. Neurology. 2018 Mar 20;90(12):e995-e1004. doi: 10.1212/WNL.0000000000005162. Epub 2018 Feb 14. PMID 29444972
- [Result] Sagris D, Papanikolaou A, Kvernland A, Korompoki E, Frontera JA, Troxel AB, Gavriatopoulou M, Milionis H, Lip GYH, Michel P, Yaghi S, Ntaios G. COVID-19 and ischemic stroke. Eur J Neurol. 2021 Nov;28(11):3826-3836. doi: 10.1111/ene.15008. Epub 2021 Jul 17. PMID 34224187
- [Result] Stein LK, Mayman NA, Dhamoon MS, Fifi JT. The emerging association between COVID-19 and acute stroke. Trends Neurosci. 2021 Jul;44(7):527-537. doi: 10.1016/j.tins.2021.03.005. Epub 2021 Apr 8. PMID 33879319
- [Result] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Result] Hingorani KS, Bhadola S, Cervantes-Arslanian AM. COVID-19 and the brain. Trends Cardiovasc Med. 2022 Aug;32(6):323-330. doi: 10.1016/j.tcm.2022.04.004. Epub 2022 Apr 21. PMID 35461991
- [Result] Cherian R, Tung ML, Chandra B. Severe COVID-19 as a virus-independent immunothrombotic process. Lancet Rheumatol. 2022 Mar;4(3):e172-e173. doi: 10.1016/S2665-9913(22)00033-9. Epub 2022 Feb 24. No abstract available. PMID 35233540
- [Result] Perico L, Benigni A, Casiraghi F, Ng LFP, Renia L, Remuzzi G. Immunity, endothelial injury and complement-induced coagulopathy in COVID-19. Nat Rev Nephrol. 2021 Jan;17(1):46-64. doi: 10.1038/s41581-020-00357-4. Epub 2020 Oct 19. PMID 33077917
- [Result] Jin Z, Liang J, Wang J, Kolattukudy PE. MCP-induced protein 1 mediates the minocycline-induced neuroprotection against cerebral ischemia/reperfusion injury in vitro and in vivo. J Neuroinflammation. 2015 Feb 27;12:39. doi: 10.1186/s12974-015-0264-1. PMID 25888869
- [Result] Tikka T, Fiebich BL, Goldsteins G, Keinanen R, Koistinaho J. Minocycline, a tetracycline derivative, is neuroprotective against excitotoxicity by inhibiting activation and proliferation of microglia. J Neurosci. 2001 Apr 15;21(8):2580-8. doi: 10.1523/JNEUROSCI.21-08-02580.2001. PMID 11306611
- [Result] Sheng Z, Liu Y, Li H, Zheng W, Xia B, Zhang X, Yong VW, Xue M. Efficacy of Minocycline in Acute Ischemic Stroke: A Systematic Review and Meta-Analysis of Rodent and Clinical Studies. Front Neurol. 2018 Dec 20;9:1103. doi: 10.3389/fneur.2018.01103. eCollection 2018. PMID 30619060
- [Result] Switzer JA, Hess DC, Ergul A, Waller JL, Machado LS, Portik-Dobos V, Pettigrew LC, Clark WM, Fagan SC. Matrix metalloproteinase-9 in an exploratory trial of intravenous minocycline for acute ischemic stroke. Stroke. 2011 Sep;42(9):2633-5. doi: 10.1161/STROKEAHA.111.618215. Epub 2011 Jul 7. PMID 21737808
- [Result] Machado LS, Sazonova IY, Kozak A, Wiley DC, El-Remessy AB, Ergul A, Hess DC, Waller JL, Fagan SC. Minocycline and tissue-type plasminogen activator for stroke: assessment of interaction potential. Stroke. 2009 Sep;40(9):3028-33. doi: 10.1161/STROKEAHA.109.556852. Epub 2009 Jul 23. PMID 19628804
- [Result] Naderi Y, Panahi Y, Barreto GE, Sahebkar A. Neuroprotective effects of minocycline on focal cerebral ischemia injury: a systematic review. Neural Regen Res. 2020 May;15(5):773-782. doi: 10.4103/1673-5374.268898. PMID 31719236
- [Result] Fagan SC, Cronic LE, Hess DC. Minocycline development for acute ischemic stroke. Transl Stroke Res. 2011 Jun 1;2(2):202-8. doi: 10.1007/s12975-011-0072-6. PMID 21909339
- [Result] Malhotra K, Chang JJ, Khunger A, Blacker D, Switzer JA, Goyal N, Hernandez AV, Pasupuleti V, Alexandrov AV, Tsivgoulis G. Minocycline for acute stroke treatment: a systematic review and meta-analysis of randomized clinical trials. J Neurol. 2018 Aug;265(8):1871-1879. doi: 10.1007/s00415-018-8935-3. Epub 2018 Jun 14. PMID 29948247
- [Derived] Lu Y, Guan L, Wu J, Yang Q, Zhang M, Zhou D, Yang H, Pan Y, Wang L, Qiu B, Liu C, Wang Y, Yang Y, Zhou X, Qu H, Liao X, Liu L, Zhao X, Bath PM, Johnston SC, Amarenco P, Turc G, Shi FD, Wang Y, Wang Y; EMPHASIS Investigators. Efficacy and safety of minocycline in patients with acute ischaemic stroke (EMPHASIS): a multicentre, double-blind, randomised controlled trial. Lancet. 2026 Jan 30:S0140-6736(25)01862-8. doi: 10.1016/S0140-6736(25)01862-8. Online ahead of print. PMID 41628627